CLINICAL TRIAL: NCT06419920
Title: Prosthetic Performance Enhancement Trial
Acronym: PROSPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: University of Washington (Other); Chapman University (Other); United States Department of Defense (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UNLV-2023-595; CDMRP-OP230011 (Other Grant/Funding Number: Department of Defence)
Record Dates: First submitted 2024-05-02; First posted 2024-05-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Amputation; Lower Limb Amputation Below Knee (Injury); Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation at Ankle (Injury); Lower Limb Amputation Knee; Lower Limb Amputation at Hip (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Feasibility study incorporating a single-blinded Phase I clinical trial with a parallel groups design, involving two treatment conditions: uneven terrain training (UT) and flat terrain (FT) training. Participants will be allocated randomly to UT and FT arms in a 6:1 ratio.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flat terrain training (Active Comparator): Walking on a standard, flat treadmill or mat.
  Interventions: Other: Flat terrain locomotor training
- Uneven terrain training (Experimental): Walking on an uneven terrain treadmill or mat.
  Interventions: Other: Uneven terrain locomotor training

INTERVENTIONS:
Other: Flat terrain locomotor training — The training will be comprised of up to 12 sets of 2-min continuous walking on a level treadmill or mat, interspersed with rest breaks of at least one minute. Training will be completed three times per week for four weeks.
  Arms: Flat terrain training
Other: Uneven terrain locomotor training — The training will be comprised of up to 12 sets of 2-min continuous walking on an uneven terrain treadmill or mat, interspersed with rest breaks of at least one minute. Training will be completed three times per week for four weeks.
  Arms: Uneven terrain training

SUMMARY:
The purpose of this research is to determine the feasibility of an uneven terrain walking program for lower limb prosthesis users. The training is designed to induce step-to-step variability during walking within a safe environment, with the aim of improving walking skill and confidence.

DETAILED DESCRIPTION:
Despite advances in the technology for artificial limbs (prostheses), falling and the fear of falling continue to be barriers to mobility for many lower limb prosthesis users after their initial rehabilitation. The loss of ability and confidence in pursuing everyday tasks negatively impacts quality of life, and ongoing physical and mental health. This study will test and improve a rehabilitation training intervention involving walking on uneven ground to improve walking skill and confidence in lower limb prosthesis users.

Lower limb prosthesis users will be recruited. Participants will be allocated randomly to receive either intervention A: training on a flat surface, or intervention B: training on an uneven surface. Depending on their ability and confidence, participants will complete the walking practice either on a treadmill or on a mat with an identical surface pattern. The walking practice will take place three times per week for four weeks. As each participant improves their ability, training tasks will be made more difficult by limiting handrail use, by increasing walking speed, and, for intervention B, also by making the walking surface more uneven.

The objectives of this pilot study are to evaluate adherence and refine the training protocols in preparation for a definitive trial that will inform rehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

* lower limb amputation at ankle (Symes) level and above
* age 18+ years
* fitted with a walking prosthesis and use it regularly for home and/or community ambulation
* good socket fit, assessed by a score of 8-10 on the socket fit comfort scale
* able to walk for three minutes at a time with or without an assistive device

Exclusion Criteria:

* leg/foot ulcer or other conditions that cause pain during weight-bearing
* poor skin integrity that could cause tissue breakdown by walking
* cardiovascular, respiratory or other critical health conditions that preclude moderate physical activity
* unilateral or bilateral upper limb absence or loss at the wrist and above that precludes use of handrails bilaterally, or would require asymmetrical adaptation to body posture for use.
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Session adherence | Through study completion, over 4 weeks
  Percentage of planned sessions attended, per participant.

SECONDARY OUTCOMES:
L-test time | Pre-intervention, within 5 days post intervention
  Time to complete L-test, in s. Participant rises from a chair and guided by cones, walks 10m forward, turns 90 degrees, walks a further 10m, turns 180 degrees, then follows the same path back to the chair and sits. Result from a single test following one practice trial is recorded.
Activities-specific Balance Confidence Scale summary score | Pre-intervention, within 5 days post intervention
  16-item self report measure recording confidence in performing activities during daily life that require balance, on numerical ratings scale, recorded as a percentage (out of 100).
Average daily activity | Pre-intervention, within 5 days post intervention
  Mean number of steps per day over 7 days, collected using ankle worn activity monitor.
Four Square Step Test time | Pre-intervention, within 5 days post intervention
  Time to complete forwards, lateral and backwards stepping pattern, in s.
Single leg stand time | Pre-intervention, within 5 days post intervention
  Time standing on one leg up to a maximum of 20s, in s.
Two-minute walk test distance | Pre-intervention, within 5 days post intervention
  Walking distance traveled in two minutes, in m.
Protocol acceptability | End of intervention week 4
  Likert scale questions and short answer questions to determine acceptability of protocol to participants, assessed qualitatively.
Recruitment feasibility - recruitment rate | From start of recruitment period, to 12 month time point.
  Number of participants recruited within one year
Recruitment feasibility - participating clinics | Through study completion, from start of recruitment period, to end of recruitment period or 30 month time point, whichever is sooner.
  Number of clinics from which at least one participant is recruited.
Recruitment feasibility - sample characteristics | Through study completion, from start of recruitment period, to end of recruitment period or 30 month time point, whichever is sooner.
  Sample characteristics of all participants enrolled in the study, regardless of completion.
Activity data evaluation | Throughout activity monitoring period, over 2 weeks
  Completeness and quality of activity monitor data, measured as number of days with valid (non-erroneous) monitoring data.
Maximum relative variability of lateral trunk velocity during uneven terrain in comparison to overground walking | Through study completion, over 4 weeks
  Medial-lateral trunk variability will be quantified during each bout of walking during each session. The maximum relative variability will be calculated as the difference in variability (standard deviation) of peak per-step lateral trunk velocity during UT walking sessions relative to that of overground walking, in m/s.
Contour depth at maximum relative variability | Through study completion, over 4 weeks
  Terrain contour depth at which the maximum relative variability was recorded, in m.
Maximum relative step width variability during uneven terrain in comparison to overground walking | Through study completion, over 4 weeks
  Step width variability will be quantified during each bout of walking during each session. The maximum relative variability will be calculated as the difference in variability (standard deviation) of step width during UT walking sessions relative to that of overground walking, in m.
Prosthesis Users Survey of Mobility t-score | Pre-intervention, within 5 days post intervention
  12-item self report tool measuring prosthesis users' mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Kent, PhD, CSci, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States